CLINICAL TRIAL: NCT00621712
Title: Clinical Assessment of a New Catheter Surface Coating With Antimicrobial Properties: Efficacy and Effect of Intensive Catheter and Exit Site Care Education
Brief Title: Clinical Assessment of a New Catheter Surface Coating With Antimicrobial Properties
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vantive Health LLC (Industry)
Collaborators: Gambro Dialysatoren GmbH (Industry); Baxter Healthcare Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Study No 2007_MBR_001; ISRCTN93939200 (Registry Identifier: ISRCTN)
Record Dates: First submitted 2008-01-31; First posted 2008-02-22 (Estimated); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Renal Insufficiency
Keywords: Renal Dialysis; Dialysis, Extracorporeal; Dialysis, Renal; Extracorporeal Dialysis
MeSH Terms: conditions — Renal Insufficiency

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Patients in group A will be provided with a commercially available and CE certified standard double lumen catheter without surface coating (GamCath® catheter, No. CE 76891).
  Interventions: Device: GamCath® central venous catheter
- B (Experimental): Patients in group B will be treated with a CE certified double lumen catheter with a new antibacterial bismuth-containing surface coating (GamCath Dolphin® Protect, No. CE 90671).
  Interventions: Device: GamCath Dolphin® Protect central venous catheter

INTERVENTIONS:
Device: GamCath® central venous catheter — choice of catheter type
  Other Names: GamCath® catheter, No. CE 76891
  Arms: A
Device: GamCath Dolphin® Protect central venous catheter — choice of catheter type
  Other Names: GamCath Dolphin® Protect, No.CE 90671
  Arms: B

SUMMARY:
The study investigates the efficacy of a catheter with antibacterial surface coating in preventing central venous catheter related infection and the effect of an intensive hygiene and catheter care education of the nursing staff on preventing central venous catheter-related infection.

DETAILED DESCRIPTION:
The risk of catheter-related bloodstream infection depends on catheter type, method and site of insertion, aseptic technique and number of manipulations. To address this problem, efforts have focused on engineering biomaterials and surfaces with antibacterial properties to prevent bacteria adhesion and biofilm formation.

In view of the necessity to reduce catheter-related bloodstream infections and of the inadequacy of currently available antimicrobially coated devices, a new antimicrobial catheter surface was developed.

Among other factors, the mode and quality of catheter handling and care of exit site is an important aspect with respect to catheter-related infections.

The clinical study aims at providing data on antimicrobial efficiency of the 2 types of CE certified double lumen catheters and a supposed additional preventive effect of intense hygiene training on catheter-related infections.

ELIGIBILITY:
Inclusion Criteria:

* central venous catheter placement
* Need for extracorporeal renal replacement therapy (acute and chronic renal failure)
* Age over 18 years
* Written informed consent
* Needed catheter length 15 cm or 20 cm

Exclusion Criteria:

* Known infectivity with Hepatitis B Virus (HBV)/Hepatitis C Virus (HCV)/Human Immunodeficiency Virus (HIV)
* Any infection associated with one or more positive blood cultures within 10 days prior to catheter implantation
* Bacteremia with a former catheter within 10 days prior to catheter implantation
* Known pregnancy
* Lactation
* Participation in another clinical study during the preceding 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2007-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Bacterial colonisation of the catheter surface | at explantation

SECONDARY OUTCOMES:
Surface deposits of thrombogenic activity | at explantation
Catheter survival | at explantation
Exit site appearance | at routine catheter care
Blood parameters | during dialysis

CONTACTS AND LOCATIONS:
Overall Officials: Christiane M Erley, Prof. Dr., Principal Investigator — St. Joseph-Krankenhaus Berlin
Locations (1):
- St. Joseph-Krankenhaus Berlin, Berlin, Germany

REFERENCES:
- [Derived] Schults JA, Kleidon T, Charles K, Young ER, Ullman AJ. Peripherally inserted central catheter design and material for reducing catheter failure and complications. Cochrane Database Syst Rev. 2024 Jun 28;6(6):CD013366. doi: 10.1002/14651858.CD013366.pub2. PMID 38940297